CLINICAL TRIAL: NCT05715164
Title: Electronic Cigarettes and Nicotine Pouches for Smoking Cessation in Pakistan: A Randomized Controlled Trial
Brief Title: Electronic Cigarettes and Nicotine Pouches for Smoking Cessation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alternative Research Initiative (Other)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Principal Investigator, Dr Abdul Hameed, Research Lead, Alternative Research Initiative
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P-0094
Record Dates: First submitted 2023-01-09; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Role of Tobacco Harm Reduction in Smoking Cessation; Efficiency and Efficacy of E-cigarettes and Nicotine Pouches; Adverse Effect of E-cigarettes and Nicotine Pouches
Keywords: E-cigarettes; Nicotine Replacement Therapy; Smoking Cessation; Tobacco Control; Tobacco Harm Reduction
MeSH Terms: conditions — Vaping; Smoking Cessation | interventions — Fluid Therapy

STUDY DESIGN:
Intervention Model Description: The baseline survey will help to evaluate the smoking status, smoking behavior, socio-demographic characteristics, health status, etc. The three-arm study design would randomize 600 participants into three groups. Of the 600 participants, 200 each will receive e-cigarettes, nicotine pouches, and basic care counseling respectively. Four basic care counseling sessions will be held over the course of 48 weeks. Every 12 weeks, a standard care counseling session will be offered, followed by a study visit to track any alterations in the user's physical or mental health as well as any side effects from using nicotine pouches or e-cigarettes. All participants will complete a follow-up survey at 60 weeks. The provision of e-cigarettes and nicotine pouches will be stopped after the first 48 weeks. The remaining 12 weeks will be without the provision of any intervention and the participants must buy these items on their own.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- E-cigarettes device plus liquid (Experimental): The 200 participants will receive e-cigarettes along with basic care counseling for 48 weeks.
  Interventions: Device: E-cigarettes device plus liquid
- Nicotine Pouches (Experimental): The 200 participants will receive nicotine pouches along with basic care counseling for 48 weeks.
  Interventions: Drug: Nicotine Pouches
- Basic care counseling about smoking cessation (Active Comparator): The 200 participants will receive basic care counseling for 48 weeks.
  Interventions: Other: Basic care counseling about smoking cessation

INTERVENTIONS:
Device: E-cigarettes device plus liquid — The four basic care counseling sessions will be held over the course of 48 weeks with the supply of e-cigarettes and liquid. Every 12 weeks, a standard care counseling session will be offered, and it will be followed by a study visit to track any alterations in the user's physical or mental health as well as any side effects from using e-cigarettes.
  Arms: E-cigarettes device plus liquid
Drug: Nicotine Pouches — The four basic care counseling sessions will be held over the course of 48 weeks with a supply of nicotine pouches. Every 12 weeks, a standard care counseling session will be offered, and it will be followed by a study visit to track any alterations in the user's physical or mental health as well as any side effects from using nicotine pouches.
  Arms: Nicotine Pouches
Other: Basic care counseling about smoking cessation — The four basic care counseling sessions will be held over the course of 48 weeks. Every 12 weeks, a standard care counseling session will be offered, and it will be followed by a study visit to track any alterations in the user's physical or mental health.
  Arms: Basic care counseling about smoking cessation

SUMMARY:
Pakistan is one of the most vulnerable low- and middle-income countries with 29 million adult active tobacco users. Smoking cessation services are lacking as the tobacco control initiatives have largely failed to address the smoking endemic. Over the last five years, Pakistan has witnessed the use of innovative tobacco harm reduction such as e-cigarettes, nicotine pouches, and non-nicotine replacement therapies (non-NRTs). However, their use remains limited.

THR products are imported legally as consumer goods and are taxable. The lack of sufficient data for THR and its application is a challenge in gauging their effectiveness in assisting smokers to quit combustible smoking. Evidence-based studies on e-cigarettes and other nicotine products are required to gauge the effectiveness of e-cigarettes and nicotine pouches as smoking cessation aids.

Keeping in view the study objectives, a sample size of 600 participants will be sufficient to assess the effectiveness of e-cigarettes and nicotine pouches for smoking cessation in Pakistan. Of these, 200 participants each will receive e-cigarettes and nicotine pouches along with basic care counseling, while the remaining 200 participants will only receive basic care counseling for 48 weeks. The association of participants' characteristics with smoking and health status will be based on bivariate and multivariate analysis. The simple t-test and variance analysis will assess the differences in intervention indicators between the control and treatment groups. For the inferential analysis, the average treatment impact of the treatments will find using quasi-experimental techniques such as difference in difference (DID) or Propensity Score Matching (PMS).

This study will be evaluated participants at baseline, after their self-decided "quit date,". The follow-up will be a survey every 12 weeks. Results may inform the public, decision-makers, and researchers about the use of e-cigarettes and nicotine pouches helping smokers to quit smoking or switch to less harmful alternatives in the short- and medium-term periods.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are at least eighteen years old.
* More than 10 combustible cigarettes smoke a day at the time of study enrollment.
* Smoked cigarettes for at least a year.
* Participants are willing to stop combustible smoking.
* Participants who can sign a written consent form.
* There can only be one applicant per household.
* Own a phone that supports text massaging.

Exclusion Criteria:

* Women who are pregnant.
* Childbearing mothers.
* Currently using other nicotine- and non-nicotine-based cessation therapies.
* Expectant ladies who intend to become pregnant during the trial's participation term.
* Experienced chest pain, or another cardiovascular event or procedure (e.g., heart attack, stroke, insertion of stent, bypass surgery).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants reported adverse events of e-cigarettes or nicotine pouches | 60 Weeks
  The primary outcome will be a long-term change in health status. The best proxy indication for demonstrating a change in tobacco smoking, which is adequate to result in a clinically relevant long-term health benefit, is unknown. In the absence of accurate health indicators, we will use the change in smoking rate from baseline and smoking cessation as primary outcomes.
Change in the number of combustible cigarettes per day | 60 Weeks
  This study will evaluate the impact of e-cigarettes and nicotine pouches on cigarettes per day (CPD) and smoking cessation (7 Day Point Abstinence) at weeks 24 and 48.
Point-prevalence abstinence | 60 Weeks
  Self-reported point-prevalence abstinence in the previous week with biochemical validation will be used exhaled carbon monoxide less than 10 parts per million (PPM).

SECONDARY OUTCOMES:
7-day point-prevalence abstinence and harm reduction | 60 Weeks
  Secondary outcomes will include 7-day point-prevalence abstinence (at all subsequent check-ups) (biochemically validated at weeks 12, 24, 36, 48, and 60). As a secondary goal, this study will analyze the harm-reduction effect of e-cigarettes and nicotine pouches, as well as the analysis of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Rawalpindi and Islamabad Centre, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hameed A, Malik D. Clinical study protocol on electronic cigarettes and nicotine pouches for smoking cessation in Pakistan: a randomized controlled trial. Trials. 2024 Jan 2;25(1):9. doi: 10.1186/s13063-023-07876-y. PMID 38167206